BERKELEY DAVIS IRVINE LOS ANGELES MERCED RIVERSIDE SAN DIEGO



SAN FRANCISCO SANTA BARBARA SANTA CRUZ

9500 GILMAN DRIVE, MC 0725 LA JOLLA, CALIFORNIA 92093-0725

HERBERT WERTHEIM SCHOOL OF PUBLIC HEALTH and HUMAN LONGEVITY SCIENCE

MyMenoPlan: Online Resource for Improving Women's Menopause Knowledge and Informed Decision-making

Principal Investigator: Andrea LaCroix, PhD
UC San Diego
Herbert Wertheim School of Public Health and Human Longevity Science
Email: alacroix@ucsd.edu

NCT: 05299983 Statistical Plan: 3/31/2023

## MyMenoPlan: Online Resource for Improving Women's Menopause Knowledge and Informed Decision-making

## **Statistical Plan**

Statistical analyses will be performed using SPSS Version 26 (IBM Corp, Armonk, NY, USA). Chi-square and F-tests will be used for comparison of frequencies and means between intervention groups.